CLINICAL TRIAL: NCT01243749
Title: Evaluation of the Endeavor Resolute Zotarolimus-Eluting Coronary Stent System in a Real-World Patient Population in China
Brief Title: RESOLUTE China Registry:
Acronym: R-C Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: IP124
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Ischemic Heart Disease; Stenotic Coronary Lesion; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease
Keywords: Target Vessel Revascularization (TVR); Target Lesion Revascularization (TLR); Myocardial Infarction (MI); Target Vessel Failure (TVF); Target Lesion Failure (TLF); Stent Thrombosis; Restenotic Lesion; Percutaneous Coronary Intervention (PCI); Real-world
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To document the safety and overall clinical performance of the Resolute Zotarolimus-Eluting Coronary Stent System in a real-world patient population requiring stent implantation.

DETAILED DESCRIPTION:
The Resolute stent is designed to support the approach of delivering drug to the coronary arterial tissue over a longer period of time than that offered by current approved DES products. This method of prolonged drug elution may address the need to control local vascular neointimal proliferation in patients with complex lesions for extended therapeutic effect. The purpose of this multi-center trial is to investigate the clinical safety and efficacy of the Endeavor Resolute drug-eluting stent in every-day patients, like stable and unstable patients with single or multi-vessel disease and/or complex lesions.

Patients should be treated according to normal hospital routine practice and in line with the applicable guidelines on percutaneous coronary interventions and the Instructions For Use of the device.

1800 patients will be enrolled from China at approximately 40 centers where Endeavor Resolute stent is commercially available.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet all of the following criteria to be eligible for treatment in the trial:

1. Age ≥ 18 years or minimum age as required by local regulations
2. The patient is an acceptable candidate for treatment with a drug-eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, the Instructions for Use of the Resolute stent and the Declaration of Helsinki
3. The patient or legal representative has been informed of the nature of the trial and has consented to participate and authorized the collection and release of his/her medical information by signing a Patient Informed Consent Form
4. Intention to electively implant at least one Resolute stent
5. The patient is willing and able to cooperate with study procedures and required follow up visits

Exclusion Criteria:

Patients will be excluded from the trial if any of the following criteria are met:

1. Known intolerance to aspirin, clopidogrel or ticlopidin, heparin, bivalirudin, cobalt, nickel, chromium, molybdenum, polymer coatings (e.g. Biolinx), zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative, or contrast media
2. Women with known pregnancy or who are lactating
3. High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
4. Currently participating in another trial that has not completed the primary endpoint or that clinically interferes with the current trial requirements
5. Planned surgery within 6 months of PCI unless dual anti-platelet therapy is maintained throughout the peri-surgical period
6. Previous enrollment in the Resolute China Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for drug-eluting stent implantation according to the applicable guidelines on percutaneous coronary interventions and the Instructions for Use of the Resolute Zotarolimus-Eluting Coronary Stent System.
  All consecutive patients eligible for drug-eluting stent implantation with the elective use of the Resolute stent in one or more target lesions are candidates to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | 12m
  Target lesion failure (TLF): a composite endpoint of cardiac death, target vessel myocardial infarction (Q wave and non-Q wave) or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods at 1 year.

SECONDARY OUTCOMES:
Overall stent thrombosis | 12m
  Overall stent thrombosis, defined as definite and probable stent thrombosis, according to the Academic Research Consortium (ARC) definition, at 1 year.
Device success, Lesion success, Procedural success | At the end of the index procedure or during hospital stay
TLF | 30 days, 6 months, 2 year, 3 year, 4 year and 5 year
  Target lesion failure (TLF): a composite endpoint of cardiac death, target vessel myocardial infarction (Q wave and non-Q wave) or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods will be assessed at 30 days, 6 months, 2 year, 3 year, 4 year and 5 year
All deaths (cardiac, vascular and non-cardiovascular) | 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
Stent thrombosis rate | at 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
  defined as definite, probable, possible, and overall stent thrombosis (according to ARC definition)
Myocardial infarction | at 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
  Q wave and non-Q wave MI
Revascularization | at 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
  target lesion and target vessel revascularization (TLR and TVR)
Significant bleeding complications and stroke | at 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
  hemorrhagic in nature
Target vessel failure (TVF) | at 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
  a composite endpoint of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization
Major adverse cardiac events (MACE) | at 30 days, 6 months, 1 year, 2 year, 3 year, 4 year and 5 year
  a composite endpoint of death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or repeat target lesion revascularization (clinically driven/clinically indicated) by percutaneous or surgical methods

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, MD, Principal Investigator — Fu Wai Hospital, Beijing, China; Jiyan Chen, MD, Principal Investigator — Guangdong Provincial People's Hospital; Lianglong Chen, MD, Principal Investigator — Fujian Medical University Union Hospital; Shaoliang Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Weimin Wang, MD, Principal Investigator — Peiking University People's Hospital; Guoying Zhu, MD, Principal Investigator — Wuhan Asia Heart Hospital
Locations (6):
- China (6):
  - Beijing Fumwai Hospital, Beijing
  - Peiking University People's Hospital, Beijing
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangdong
  - Nanjing First Hospital, Nanjing
  - Wuhan Asia Heart Hospital, Wuhan

REFERENCES:
- [Result] Qiao S, Chen L, Chen S, Wang W, Zhu G. One-year outcomes from an all-comers chinese population of patients implanted with the resolute zotarolimus-eluting stent. Am J Cardiol. 2014 Feb 15;113(4):613-20. doi: 10.1016/j.amjcard.2013.10.042. Epub 2013 Nov 23. PMID 24365120